CLINICAL TRIAL: NCT03123939
Title: Phase IIIb Study for Relapsed/Refractory Pediatric/Young Adult Acute Lymphoblastic Leukemia Patients to be Treated With CTL019
Brief Title: Phase III B in Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019B2001X; 2016-001991-31 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; Acute Lymphoblastic Leukemia; CTL019; relapsed/refractory pediatric/young adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CTL019 (Experimental): CTL019 transduced T cells were given as a single dose of 0.2 to 5.0 × 10^6 autologous CTL019 transduced viable T cells per kg body weight (for patients ≤ 50 kg) and 0.1 to 2.5 × 10^8 CTL019 transduced viable T cells (for patients > 50 kg)
  Interventions: Biological: CTL019

INTERVENTIONS:
Biological: CTL019 — CTL019 transduced T cells were given as a single dose of 0.2 to 5.0 × 10^6 autologous CTL019 transduced viable T cells per kg body weight (for patients ≤ 50 kg) and 0.1 to 2.5 × 10^8 CTL019 transduced viable T cells (for patients > 50 kg)

SUMMARY:
This is a single arm, open-label, multi-center, phase III B study to determine the safety and efficacy of CTL019 in pediatric/young adult patients with r/r B-cell Acute Lymphoblastic Leukemia (ALL).

DETAILED DESCRIPTION:
This was a single-arm, multi-centeric Phase IIIb study provided pediatric/young adult patients with r/r B-cell ALL the opportunity to be treated with CTL019. The main purpose of this study was to assess the safety of CTL019 for up to 12 months after the CTL019 infusion. The study had the following sequential phases for all patients: Screening including leukapheresis, Pre-Treatment (Cell Product Preparation and Lymphodepleting Chemotherapy), Treatment and Follow-up, and Long-Term Follow-Up (LTFU). The end of study (EOS) was defined as the last patient's last visit, which was the last patient's Month 12 evaluation, or the time of premature withdrawal. All patients were followed in this study for up to 12 months after the CTL019 infusion.

ELIGIBILITY:
Inclusion Criteria:

Relapsed or refractory B-cell ALL in pediatric or young adult patients:

1. Second or greater bone marrow relapse.
2. Any bone marrow relapse after allogeneic SCT and must be ≥ 4 months from SCT at the time of CTL019 infusion OR
3. Primary refractory as defined by not achieving a CR after 2 cycles of a standard chemotherapy regimen or chemorefractory as defined by not achieving a CR after 1 cycle of standard chemotherapy for relapsed leukemia OR
4. Patients with Philadelphia chromosome positive (Ph+) ALL are eligible if they are intolerant to or have failed 2 lines of tyrosine kinase inhibitor (TKI) therapy, or if TKI therapy is contraindicated OR
5. Ineligible for allogeneic SCT

For relapsed patients, CD19 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry within 3 months of program entry.For relapsed or refractory patients previously treated with blinatumomab, CD19 tumor expression must be demonstrated (via flow cytometry) at Screening.

Adequate organ function defined as:

1. A serum creatinine based on age/gender as follows: Maximum Serum Creatinine (mg/dL). Age Male Female: to < 2 years 0.6 0.6; to < 6 years 0.8 0.8; 6 to < 10 years 1.0 1.0; 10 to < 13 years 1.2 1.2; 13 to < 16 years 1.5 1.4; ≥ 16 years 1.7 1.4.
2. ALT ≤ 5 times the upper limit of normal (ULN) for age.
3. Bilirubin < 2.0 mg/dL.
4. Minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air.
5. Left Ventricular Shortening Fraction ≥ 28% by echocardiogram, or Left Ventricular Ejection Fraction ≥ 45% by echocardiogram or Multiple Uptake Gated Acquisition (MUGA).

Life expectancy > 12 weeks.

Age less than 26 at the time of screening.

Karnofsky (age ≥16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening.

Patients previously treated with blinatumomab who have detectable leukemia and documented CD19+ expression (via flow cytometry) and confirmed absence of CD19- leukemic blasts at Screening may be included. In this case, at least 1 week washout period must be applied from last dose of blinatumomab to start of leukapheresis. Patients previously treated with blinatumomab with no detectable MRD (i.e. MRD negative demonstrated by leukemic blasts < 0.01%) will be excluded.

Must have a leukapheresis product of non-mobilized cells received and accepted by the manufacturing site.

Patients with active CNS leukemia involvement defined as CNS-3 by CSF findings only are eligible but will have their CTL019 infusion delayed until CNS disease is reduced to CNS-1 or CNS-2 by CSF findings. Patients with other forms of active CNS-3 leukemic involvement such as CNS parenchymal or ocular disease, cranial nerve involvement or significant leptomeningeal disease are not eligible. However, such patients with other forms of CNS-3 leukemic involvement (non-CSF involvement) are eligible if there is documented evidence of disease stabilization for at least 3 months prior to CTL019 infusion. Patients must have no acute/ongoing neurologic toxicity > Grade 1 with the exception of a history of controlled seizures or fixed neurologic deficits that have been stable/improving over the past 3 months.

Exclusion criteria Isolated extra-medullary disease relapse. Concomitant genetic syndromes associated with bone marrow failure states: Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Patients with Down Syndrome will not be excluded.

Patients with Burkitt's lymphoma/leukemia (i.e. patients with mature B-cell ALL, leukemia with B-cell surface immunoglobulin (sIg) positive and kappa or lambda restricted positivity ALL, with FAB L3 morphology and /or a MYC translocation).

Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease.

Prior treatment with any gene therapy product. Prior treatment with any anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy, except for patients pre-treated with blinatumomab Active or latent hepatitis B or active hepatitis C (test within 8 weeks of screening), or any uncontrolled infection at screening Human immunodeficiency virus (HIV) positive test within 8 weeks of screening. Presence of grade 2 to 4 acute or extensive chronic GVHD. Uncontrolled acute life threatening bacterial, viral or fungal infection at Screening Investigational medicinal product within the last 30 days prior to screening. Pregnant or nursing women.Women of child-bearing potential and all male participants, unless they are using highly effective methods of contraception for a period of 1 year after the CTL019 infusion.

The following medications are excluded:

1. Steroids: Therapeutic systemic doses of steroids must be stopped > 72 hours prior to CTL019 infusion.
2. Allogeneic cellular therapy: Any donor lymphocyte infusions must be completed > 6 weeks prior to CTL019 infusion.
3. GVHD therapies: Any systemic drug used for GVHD must be stopped > 4 weeks prior to CTL019 infusion to confirm that GVHD recurrence is not observed.
4. Chemotherapy:

   * TKIs and hydroxyurea must be stopped > 72 hours prior to CTL019 infusion.
   * must be stopped > 1 week prior to CTL019 infusion: vincristine, 6-mercaptopurine, 6-thioguanine, methotrexate < 25 mg/m2, cytosine arabinoside < 100 mg/m2/day, asparaginase (non pegylated).
   * must be stopped > 2 weeks prior to CTL019 infusion: salvage chemotherapy (e.g. clofarabine, cytosine arabinoside > 100 mg/m2, anthracyclines, cyclophosphamide, methotrexate ≥ 25 mg/m2).
   * Pegylated-asparaginase must be stopped > 4 weeks prior to CTL019 infusion.
5. CNS disease prophylaxis: CNS prophylaxis treatment must be stopped > 1 week prior to CTL019 infusion (e.g. intrathecal methotrexate).
6. Radiotherapy

   * Non-CNS site of radiation must be completed > 2 weeks prior to CTL019 infusion.
   * CNS directed radiation must be completed > 8 weeks prior to CTL019 infusion.
7. Anti T-cell antibodies: Administration of any T cell lytic or toxic antibody (e.g. alemtuzumab) within 8 weeks prior to CTL019 is prohibited Other protocol-defined inclusion/exclusion may apply

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Ghent, Belgium
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Frankfurt, Germany
- Novartis Investigative Site, Monza, MB, Italy
- Novartis Investigative Site, Kyoto, Japan
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Laetsch TW, Maude SL, Balduzzi A, Rives S, Bittencourt H, Boyer MW, Buechner J, De Moerloose B, Qayed M, Phillips CL, Pulsipher MA, Hiramatsu H, Tiwari R, Grupp SA. Tisagenlecleucel in pediatric and young adult patients with Down syndrome-associated relapsed/refractory acute lymphoblastic leukemia. Leukemia. 2022 Jun;36(6):1508-1515. doi: 10.1038/s41375-022-01550-z. Epub 2022 Apr 14. PMID 35422096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 11 study centers across 9 countries (Austria, Belgium, Canada, Germany, Spain, France, Italy, Japan, Norway).
Pre-assignment Details: This was a single arm study.
Period: Overall Study
Arm/Group | CTL019
Started (enrolled participants) | 74
CTL019 Infused (all enrolled participants who received CTL019 infusion) | 69
Full Analysis Set (FAS) (all enrolled participants who received CTL019 infusion) | 69
Cellular Kinetic Analysis Set (CKAS) (participants who had at least 1 sample providing evaluable data) | 69
Safety Set (SAF) (all enrolled participants who received CTL019 infusion) | 69
Completed | 33
Not Completed | 41
Not completed — Lack of Efficacy | 6
Not completed — Death | 5
Not completed — Physician Decision | 2
Not completed — Subject/guardian decision | 2
Not completed — Lost to Follow-up | 1
Not completed — New therapy for study indication | 1
Not completed — Protocol deviation | 1
Not completed — Progressive disease | 18
Not completed — Discontinued prior to CTL019 infusion due to death | 4
Not completed — Discontinued prior to CTL019 infusion due to technical problems | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Arm/Group | CTL019
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 52
  Black or African American | 2
  Asian | 4
  American Indian or Alaska Native | 1
  Unknown | 3
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse events were collected from CTL019 infusion until end of study, up to 12 months
Time Frame: From CTL019 infusion until end of study, up to 12 months
Population: The Safety Set (SAF) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants | 69

2. Secondary Outcome: Overall Remission Rate (ORR)
Description: ORR is defined as the proportion of participants with a best overall disease response of Complete remission (CR) or CR with incomplete blood count recovery (CRi), where the best overall disease response is defined as the best disease response recorded from CTL019 infusion until Month 6.
Time Frame: From CTL019 infusion until Month 6
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants | 57

3. Secondary Outcome: Number of Participants Who Achieved CR or CRi at Month 6 Without Stem Cell Transplantation (SCT)
Description: Proportion of participants who achieved CR or CRi at Month 6 without stem cell transplantation between CTL019 infusion and Month 6 response assessment
Time Frame: Month 6
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants | 41

4. Secondary Outcome: Number of Participants Who Achieved CR or CRi and Then Proceeded to Stem Cell Transplantation (SCT) While in Remission Before Month 6 Assessment
Description: Proportion of participants who achieved CR or CRi and then proceeded to stem cell transplantation while in remission prior to Month 6 response assessment.
Time Frame: From CTL019 infusion until Month 6
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants | 1

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the duration of remission from the date when the response criteria of CR or CRi was first met post CTL019 infusion to the date of relapse or death due to acute lymphoblastic leukemia (ALL), whichever occured first.
Time Frame: Actual reported Time Frame: up to 14.4 months post CTL019 infusion (planned follow-up period per protocol was only 12 months post CTL019 infusion)
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019 and had a best overall response of CR or CRi
Measure: Median (Full Range); unit: Months
Arm/Group | CTL019
Number analyzed (Participants) | 57
Months | 8.9 [1.7 to 14.4]

6. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS is measured by the time from achievement of CR or CRi whichever occured first post CTL019 infusion, to relapse or death due to any cause during CR or CRi.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | CTL019
Number analyzed (Participants) | 57
Months | 8.9 [1.7 to 14.4]

7. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is the time from date of CTL019 infusion to the earliest of death, relapse or treatment failure.
Time Frame: Actual reported Time Frame: up to 15.1 months post CTL019 infusion (planned follow-up period per protocol was only 12 months post CTL019 infusion)
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Median (Full Range); unit: Months
Arm/Group | CTL019
Number analyzed (Participants) | 69
Months | 8.97 [0.0 to 15.1]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from date of CTL019 infusion to the date of death due to any reason
Time Frame: Actual reported Time Frame: up to 24.4 months post CTL019 infusion (planned follow-up period per protocol was only 12 months post CTL019 infusion)
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Median (Full Range); unit: Months
Arm/Group | CTL019
Number analyzed (Participants) | 69
Months | 11.7 [0.3 to 24.4]

9. Secondary Outcome: Number of Participants Who Attained CR or CRi at Day 28
Description: Proportion of participants who attained CR or CRi at Day 28 post CTL019 infusion.
Time Frame: Day 28
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants | 59

10. Secondary Outcome: Number of Participants Who Attained CR or CRi at Day 28 by Baseline Bone Marrow Tumor Burden
Description: Proportion of participants who attained CR or CRi at Day 28 post CTL019 infusion by baseline bone marrow tumor burden.
Time Frame: Day 28
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019 and had a baseline bone marrow tumor burden result
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 66
Participants
  Low tumor burden (morphologic result < 50%) | 26
  High tumor burden (morphologic result ≥ 50%) | 40

11. Secondary Outcome: Bone Marrow Minimum Residual Disease (MRD) Status by Flow Cytometry on Day 28 Post CTL019 Infusion
Description: MRD in ALL refers to the presence of leukemic cells below the threshold of detection using conventional morphologic methods. The most frequently used methods for MRD assessment include multicolor flow cytometry to detect abnormal immunophenotypes and polymerase chain reaction (PCR) assays to detect clonal rearrangements in immunoglobulin heavy chain genes and/or T-cell receptor genes or fusion transcripts (e.g. BCR-ABL (Philadelphia chromosome)). The results include the descriptive summary of MRD qualitative result (positive/negative) before treatment and at Day 28 after treatment and before HSCT by local assessment (flow cytometry).
Time Frame: Enrollment/Pre-chemotherapy and Day 28
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants
  Enrollment/Pre-Chemotherapy: Negative | 0
  Enrollment/Pre-Chemotherapy: Positive | 51
  Enrollment/Pre-Chemotherapy: Unknown | 4
  Enrollment/Pre-Chemotherapy: Not done | 1
  Enrollment/Pre-Chemotherapy: Missing | 13
  Day 28: Negative | 44
  Day 28: Positive | 4
  Day 28: Unknown | 2
  Day 28: Not done | 0
  Day 28: Missing | 19

12. Secondary Outcome: Bone Marrow Minimum Residual Disease (MRD) Status by qPCR on Day 28 Post CTL019 Infusion
Description: MRD in ALL refers to the presence of leukemic cells below the threshold of detection using conventional morphologic methods. The most frequently used methods for MRD assessment include multicolor flow cytometry to detect abnormal immunophenotypes and polymerase chain reaction (PCR) assays to detect clonal rearrangements in immunoglobulin heavy chain genes and/or T-cell receptor genes or fusion transcripts (e.g. BCR-ABL (Philadelphia chromosome)). The results include the descriptive summary of MRD qualitative result (positive/negative) before treatment and at Day 28 after treatment and before HSCT by local assessment (qPCR).
Time Frame: Enrollment/Pre-chemotherapy and Day 28
Population: Full Analysis Set (FAS) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants
  Enrollment/Pre-Chemotherapy: Negative | 1
  Enrollment/Pre-Chemotherapy: Positive | 32
  Enrollment/Pre-Chemotherapy: Unknown | 4
  Enrollment/Pre-Chemotherapy: Not done | 0
  Enrollment/Pre-Chemotherapy: Missing | 32
  Day 28: Negative | 31
  Day 28: Positive | 3
  Day 28: Unknown | 0
  Day 28: Not done | 0
  Day 28: Missing | 35

13. Secondary Outcome: Incidence of Immunogenicity Against CTL019 - Humoral Immunogenicity
Description: The humoral immunogenicity assessment included evaluation of pre-existing (pre-treatment) and post-treatment anti-CTL019 antibodies to examine the incidence of immunogenicity with treatment.
Time Frame: Baseline, Day 14, Day 28, Month 3, Month 6 and Month 12
Population: The Safety Set (SAF) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants
  Baseline: Positive | 62
  Baseline: Negative | 7
  Baseline: Missing | 0
  Day 14: Positive | 53
  Day 14: Negative | 14
  Day 14: Missing | 2
  Day 28: Positive | 50
  Day 28: Negative | 13
  Day 28: Missing | 6
  Month 3: Positive | 53
  Month 3: Negative | 5
  Month 3: Missing | 11
  Month 6: Positive | 44
  Month 6: Negative | 4
  Month 6: Missing | 21
  Month 12: Positive | 32
  Month 12: Negative | 1
  Month 12: Missing | 36

14. Secondary Outcome: Incidence of Immunogenicity Against CTL019 - Cellular Immunogenicity
Description: The cellular immunogenicity assessment included percentage of CD4+ and CD8+ T- cells specific for CTL019.
Time Frame: Baseline, Day 14, Day 28, Month 3, Month 6 and Month 12
Population: The Safety Set (SAF) comprised of all the participants who received an infusion of CTL019
Measure: Count of Participants; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 69
Participants
  CTL019 Pool 1 CD3+ CD4+ IFNg+ Baseline | 69
  CTL019 Pool 1 CD3+ CD4+ IFNg+ Day 14 | 65
  CTL019 Pool 1 CD3+ CD4+ IFNg+ Day 28 | 63
  CTL019 Pool 1 CD3+ CD4+ IFNg+ Month 3 | 58
  CTL019 Pool 1 CD3+ CD4+ IFNg+ Month 6 | 51
  CTL019 Pool 1 CD3+ CD4+ IFNg+ Month 12 | 34
  CTL019 Pool 2 CD3+ CD4+ IFNg+ Baseline | 69
  CTL019 Pool 2 CD3+ CD4+ IFNg+ Day 14 | 65
  CTL019 Pool 2 CD3+ CD4+ IFNg+ Day 28 | 63
  CTL019 Pool 2 CD3+ CD4+ IFNg+ Month 3 | 58
  CTL019 Pool 2 CD3+ CD4+ IFNg+ Month 6 | 51
  CTL019 Pool 2 CD3+ CD4+ IFNg+ Month 12 | 34
  CTL019 Pool 1 CD3+ CD8+ IFNg+ Baseline | 69
  CTL019 Pool 1 CD3+ CD8+ IFNg+ Day 14 | 65
  CTL019 Pool 1 CD3+ CD8+ IFNg+ Day 28 | 63
  CTL019 Pool 1 CD3+ CD8+ IFNg+ Month 3 | 58
  CTL019 Pool 1 CD3+ CD8+ IFNg+ Month 6 | 51
  CTL019 Pool 1 CD3+ CD8+ IFNg+ Month 12 | 34
  CTL019 Pool 2 CD3+ CD8+ IFNg+ Baseline | 69
  CTL019 Pool 2 CD3+ CD8+ IFNg+ Day 14 | 65
  CTL019 Pool 2 CD3+ CD8+ IFNg+ Day 28 | 63
  CTL019 Pool 2 CD3+ CD8+ IFNg+ Month 3 | 58
  CTL019 Pool 2 CD3+ CD8+ IFNg+ Month 6 | 51
  CTL019 Pool 2 CD3+ CD8+ IFNg+ Month 12 | 34

15. Secondary Outcome: AUC0-28d: PK Parameters for CTL019 by qPCR
Description: Area under the concentration-time curve of CTL019 in the peripheral blood after single dose administration from time zero to Day 28 after single dose administration as measured by qPCR.
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28
Population: Cellular kinetic analysis set (CKAS) consisted of participants in the FAS who had at least 1 sample providing evaluable cellular kinetic data and had non-missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug*day
Arm/Group | CTL019
Number analyzed (Participants) | 57
copies/ug*day | 365000 (174.5)

16. Secondary Outcome: AUC0-84d: PK Parameters for CTL019 by qPCR
Description: Area under the concentration-time curve of CTL019 in the peripheral blood after single dose administration from time zero to Day 84 after single dose administration as measured by qPCR.
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28 and 84
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies/ug*day
Arm/Group | CTL019
Number analyzed (Participants) | 46
Copies/ug*day | 555000 (193.3)

17. Secondary Outcome: Cmax: PK Parameters for CTL019 by qPCR
Description: The maximum (peak) observed in peripheral blood drug concentration after single dose administration
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28, Month 3, 6, 9 and 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | CTL019
Number analyzed (Participants) | 62
copies/ug | 35300 (215.7)

18. Secondary Outcome: Clast: PK Parameters for CTL019 by qPCR
Description: The last observed in peripheral blood drug concentration after single dose administration.
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28, Month 3, 6, 9 and 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | CTL019
Number analyzed (Participants) | 62
copies/ug | 240 (147.3)

19. Secondary Outcome: Tmax: PK Parameters for CTL019 by qPCR
Description: The time to reach maximum (peak) peripheral blood drug concentration after single dose administration.
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28, Month 3, 6, 9 and 12
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | CTL019
Number analyzed (Participants) | 62
days | 10.0 [5.86 to 17.5]

20. Secondary Outcome: T1/2: PK Parameters for CTL019 by qPCR
Description: The half-life associated with the elimination phase slope of a semi logarithmic concentration-time curve (days) in peripheral blood.
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28, Month 3, 6, 9 and 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | CTL019
Number analyzed (Participants) | 35
days | 63.8 (182.1)

21. Secondary Outcome: Tlast: PK Parameters for CTL019 by qPCR
Description: The time to reach the last observed quantifiable concentration in peripheral blood after single dose administration.
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28, Month 3, 6, 9 and 12
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | CTL019
Number analyzed (Participants) | 62
days | 269 [12.9 to 379]

22. Secondary Outcome: AUC0-28d by Maximum Cytokine Release Syndrome (CRS) Grade
Description: AUC0-28d from time zero to Day 28 after single dose administration as measured by qPCR. PK results were presented by the maximum Penn Grading Scale (Grade 1 to 4):
  1. - Mild reaction
  2. - Moderate reaction
  3. - More severe reaction
  4. - Life-threatening complications
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug*day
Arm/Group | CTL019
Number analyzed (Participants) | 57
copies/ug*day
  No CRS: number analyzed (Participants) | 17
  No CRS | 141000 (130.6)
  Grade 1/2: number analyzed (Participants) | 19
  Grade 1/2 | 374000 (72.6)
  Grade 3: number analyzed (Participants) | 9
  Grade 3 | 643000 (272.8)
  Grade 4: number analyzed (Participants) | 12
  Grade 4 | 890000 (119.1)

23. Secondary Outcome: Cmax by Maximum Cytokine Release Syndrome (CRS) Grade
Description: The maximum (peak) observed in peripheral blood drug concentration after single dose administration. PK results were presented by the maximum Penn Grading Scale (Grade 1 to 4):
  1. - Mild reaction
  2. - Moderate reaction
  3. - More severe reaction
  4. - Life-threatening complications
Time Frame: Day 1 10 min post-infusion, Day 4, 7, 11, 14, 28, Month 3, 6, 9 and 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/ug
Arm/Group | CTL019
Number analyzed (Participants) | 62
copies/ug
  No CRS: number analyzed (Participants) | 18
  No CRS | 16300 (157.8)
  Grade 1/2: number analyzed (Participants) | 23
  Grade 1/2 | 31200 (199.3)
  Grade 3: number analyzed (Participants) | 9
  Grade 3 | 66600 (299.9)
  Grade 4: number analyzed (Participants) | 12
  Grade 4 | 87900 (84.9)

24. Post Hoc Outcome: Total Number of Deaths
Description: Deaths were reported in the pre-treatment period (without receiving a CTL019 infusion) and post-treatment period (after receiving a CTL019 infusion).
Time Frame: Pre-treatment period: up to 81 days post signed informed consent; Post-treatment period: up to 24.4 months post CTL019 infusion (planned follow-up period per protocol was only 12 months post CTL019 infusion)
Population: all enrolled participants
Measure: Number; unit: Participants
Arm/Group | CTL019
Number analyzed (Participants) | 74
Participants
  Pre-treatment (without CTL019 infusion) | 4
  Post-treatment: ≤30 days (after CTL019 infusion): number analyzed (Participants) | 69
  Post-treatment: ≤30 days (after CTL019 infusion) | 4
  Post-treatment: >30 days (after CTL019 infusion): number analyzed (Participants) | 69
  Post-treatment: >30 days (after CTL019 infusion) | 5

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from CTL019 infusion, until approximately 12 months post infusion. For all-cause mortality, the data are presented from CTL019 infusion up to 24.4 months post infusion.
Description: Any signs or symptoms that occurred from CTL019 infusion until end of study.
Groups:
- All Subjects - CTL019: CTL019 transduced T cells were given as a single dose of 0.2 to 5.0 × 10^6 autologous CTL019 transduced viable T cells per kg body weight (for patients ≤ 50 kg) and 0.1 to 2.5 × 10^8 CTL019 transduced viable T cells (for patients > 50 kg)
Arm/Group | All Subjects - CTL019
All-Cause Mortality (participants affected / at risk) | 9/69
Serious Adverse Events (participants affected / at risk) | 50/69
Other Adverse Events (participants affected / at risk) | 66/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects - CTL019 (N=69)
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 11
Hepatocellular injury (Hepatobiliary disorders) | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Cytokine release syndrome (Immune system disorders) | 28
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1
Alternaria infection (Infections and infestations) | 1
Aspergillus infection (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 2
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cellulitis orbital (Infections and infestations) | 1
Central nervous system infection (Infections and infestations) | 1
Cerebral fungal infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia haemophilus (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Splinter (Injury, poisoning and procedural complications) | 1
Blood fibrinogen decreased (Investigations) | 1
Chest X-ray abnormal (Investigations) | 1
Immunoglobulins decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Facial paralysis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects - CTL019 (N=69)
Anaemia (Blood and lymphatic system disorders) | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Sinus tachycardia (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Chills (General disorders) | 4
Face oedema (General disorders) | 6
Fatigue (General disorders) | 7
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 5
Pyrexia (General disorders) | 24
Allergy to immunoglobulin therapy (Immune system disorders) | 4
Cytokine release syndrome (Immune system disorders) | 30
Hypogammaglobulinaemia (Immune system disorders) | 21
Nasopharyngitis (Infections and infestations) | 9
Rhinitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 8
Blood fibrinogen decreased (Investigations) | 4
Immunoglobulins decreased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 10
White blood cell count decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 16
Seizure (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 5
Haematuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 6
Petechiae (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 10
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03123939/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT03123939/SAP_001.pdf